CLINICAL TRIAL: NCT01558726
Title: Effectiveness of Case Management for Crack Users Who Seek Treatment in CAPSad in Six Brazilian Capitals
Brief Title: Case Management for Crack Users Who Seek Treatment in CAPSad in Brazil
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Rio Grande do Sul (Other)
Collaborators: Hospital de Clinicas de Porto Alegre (Other); Brazilian Secretariat for Drug Policies (SENAD) (Unknown); Federal University of Bahia (Other); Federal University of Espirito Santo (Other); Universidade Federal do Rio de Janeiro (Other); Faculdade de Medicina do ABC (Other); University of Brasilia (Other)
Responsible Party: Principal Investigator, Professor Flavio Pechansky, Director of Center for Drug and Alcohol Research (CPAD-UFRGS), Federal University of Rio Grande do Sul
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10-0176
Record Dates: First submitted 2012-03-17; First posted 2012-03-20 (Estimated); Last update posted 2012-03-20 (Estimated); Status verified 2012-03

CONDITIONS: Crack Abuse or Dependence
Keywords: Case Management; Crack abuse/dependents; Evaluation; Inpatient; ASI; Treatment retention; Abstinence
MeSH Terms: interventions — Case Management

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Case management (Experimental)
  Interventions: Behavioral: Case Management (Strength-Based)
- Usual treatment (Active Comparator): Usual treatment of the CAPSad
  Interventions: Behavioral: Usual Treatment

INTERVENTIONS:
Behavioral: Case Management (Strength-Based) — To improve the cases sharing between CAPSad and other health institutions and individuals and increase the strengths of the patient to cope with problems related to the crack use.
  Arms: Case management
Behavioral: Usual Treatment — The usual treatment used for regular patients of CAPSad
  Arms: Usual treatment

SUMMARY:
The purpose of this study is to evaluate the effectiveness of a Case Management (CM) intervention in crack users applied in Psychosocial Care Centers - Alcohol and Drugs (CAPSad) by trained social workers, in comparison to CAPSad conventional treatment on 30 and 90 days, considering the following outcomes: treatment retention, abstinence and changes in severity scores of the sixth version of Addiction Severity Index (ASI6) scale. The study hypothesis are: 1) The CM is going to improve the retention of crack users (cases) during the 3-month follow-up compared with usual care (controls); 2)Individuals who received the intervention with GC are going to present a higher rate of abstinence; 3)The summary scores of the ASI6 will be significantly lower in cases than in controls, at the end of 3 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of crack abuse or dependence
* > 18 years old
* Initiating treatment (maximum of 1 month)

Exclusion Criteria:

* Homeless without permanent contact
* Psychotic symptoms during the intake interview

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2011-10; Primary Completion 2012-08 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
Treatment retention | 3 months

SECONDARY OUTCOMES:
Crack abstinence | 3 months
ASI subareas scores | 3 months
  ASI (Addiction Severity Index)

CONTACTS AND LOCATIONS:
Overall Officials: Flavio Pechansky, PhD, Principal Investigator — Center for Drug and Alcohol Research (CPAD) of Federal University of Rio Grande do Sul
Locations (1):
- Center for Drug and Alcohol Research (CPAD) of Federal University of Rio Grande do Sul (UFRGS), Porto Alegre, Rio Grande do Sul, Brazil